CLINICAL TRIAL: NCT04429919
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of AP-325 in Subjects With Peripheral Post-surgical Neuropathic Pain
Brief Title: AP-325 in Subjects With Peripheral Post-surgical Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Algiax Pharmaceuticals GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-325.04
Record Dates: First submitted 2020-05-29; First posted 2020-06-12 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Post-surgical Neuropathic Pain
Keywords: AP-325; Phase IIa; PPNP; post-surgical neuropathic pain

STUDY DESIGN:
Intervention Model Description: placebo controlled, Phase IIa clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AP-325 (Experimental): 25 mg capsule for oral use, 4 capsules (100 mg) once daily in the morning before meals
  Interventions: Drug: AP-325
- Placebo (Placebo Comparator): 4 capsules once daily in the morning before meals
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AP-325 — During the 10-day double-blind treatment period (Days 1 to 10), subjects will take 4 capsules of the IMP orally once daily in the morning before breakfast.
  Arms: AP-325
Drug: Placebo — During the 10-day double-blind treatment period (Days 1 to 10), subjects will take 4 capsules of the IMP orally once daily in the morning before breakfast.
  Arms: Placebo

SUMMARY:
This is a Phase IIa randomized, double-blind, placebo-controlled study. The study objective is to investigate the efficacy and safety of repeat oral dosing of the investigational medicinal product (IMP) AP-325 for the treatment of peripheral post-surgical neuropathic pain (PPNP) after breast surgery (breast-conserving surgery, mastectomy, surgery to remove lymph nodes), chest surgery (e.g. thoracotomy, video assisted thoracoscopy and sternotomy), hernia repair of the abdominal wall (e.g. femoral hernia repairs, inguinal hernia repairs, umbilical hernia repair or incisional hernia repair), abdominal surgery (e.g. cholecystectomy, appendectomy but also see exclusion criterion 15), varicose vein surgery or gynecologic surgery (e.g. hysterectomy, C-section).

DETAILED DESCRIPTION:
This is a Phase IIa randomized, double-blind, placebo controlled, parallel group study to evaluate the efficacy (by changes in Pain Intensity Numerical Rating Scale [PI-NRS]) and safety (by monitoring adverse events) of AP-325 in subjects with PPNP.

The clinical trial will be conducted in Germany, Spain, Czech Republic, Belgium and France.

Eligible subjects will undergo a 2-week run-in period consisting of a washout-period of prohibited medications in the 1st week and a baseline period in the 2nd week. If subjects have at least 5 self-reported pain assessments in the baseline period (documented in a diary) and meet the required pain criteria, they will be randomized to AP-325 or placebo in a 1:1 ratio.

Subjects will take the IMP (AP-325 or placebo) for 10 days (double-blind treatment period; Days 1-10) and then be followed up for a further 26 days (drug-free period; Days 11-36). An end of study visit will be performed on Day 36.

At least 96 subjects (48 for each treatment) need to be analyzed for the primary endpoint at Day 10 to reach the power estimate (120 subjects should be screened for the study).

AP-325 100 mg (4 x 25 mg capsules) or Placebo (4 capsules) will be orally taken once daily in the morning before meals for 10 consecutive days.

Pain will be assessed, and quality of life will be investigated using standardized and validated questionnaires [Pain Intensity Numerical Rating Scale (PI-NRS), patient global impression of change (PGIC), neuropathic pain symptom inventory (NPSI) questionnaire, daily sleep interference scale (DSIS) score, hospital anxiety and depression scale (HADS)].

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years and not older than 80 years
2. Subjects with a diagnosis of chronic post-surgical neuropathic pain after breast surgery (e.g. breast-conserving surgery, mastectomy, surgery to remove lymph nodes), chest surgery (e.g. thoracotomy, video assisted thoracoscopy and sternotomy), hernia repair of the abdominal wall (e.g. femoral hernia repairs, inguinal hernia repairs, umbilical hernia repair or incisional hernia repair), abdominal surgery (e.g. cholecystectomy, appendectomy but also see exclusion criterion 15), varicose vein surgery or gynecologic surgery (e.g. hysterectomy, C-section)
3. The chronic post-surgical pain developed or increased in intensity after the surgical procedure and persisted beyond the healing process, i.e. at least 3 months after the initiating event, as defined according to the international association for the study of pain (IASP) classification of chronic pain for ICD-11 (Schug et al., 2019)
4. Subjects must have 'probable' or 'definite' neuropathic pain as assessed by the revised IASP special interest group on neuropathic pain (NeuPSIG) grading system (Finnerup et al., 2016)
5. Subjects must be willing and able to discontinue and washout prohibited substances including

   * pain medications (e.g. antidepressants, anticonvulsants/antiepileptics, selective serotonin and dual reuptake inhibitors, opioids, long-acting benzodiazepines, muscle relaxants, and topical analgesics), except the rescue medication, and
   * substances known to be inhibitors or inducers of CYP2C9 and inhibitors of CYP3A4 for specific washout periods of at least 5 times the drug half-life Note: Subjects using prohibited substances for other indications than neuropathic pain, e.g. antiepileptics for the treatment of epilepsy, may not be included in the study, because a discontinuation of such medication is not medically justifiable.
6. Permitted concomitant medications must have been stable for at least 4 weeks prior to Day -14 and any non-pharmacological therapies (e.g. physiotherapy, acupuncture and transcutaneous electrical neural stimulation) must have been initiated at least 3 weeks prior to Screening
7. Female subjects must not be pregnant or breastfeeding and be

   * of non-childbearing potential or
   * if of childbearing potential, use a highly effective contraceptive method from start of the IMP intake until 30 days after the last IMP intake and have a negative pregnancy test at Screening (blood test)
8. Male subjects must agree, from start of the IMP intake until 3 months after the last IMP intake, to refrain from donating sperm and use a male condom when having sexual intercourse with a woman of childbearing potential at any time and advise her to use a highly effective contraceptive method
9. Subjects must understand the nature of the study procedures and provide written informed consent prior to any study-related procedures
10. Body weight ≥55 kg for men and ≥50 kg for women
11. Body mass index (BMI) <40 kg/m²

Exclusion Criteria:

1. Subjects with neuropathic pain not a result of a surgical procedure as defined in inclusion criterion 2
2. Subjects with any other coexisting pain that cannot be discriminated from post-surgical neuropathic pain, in the opinion of the subject or clinician e.g., the pain is at least partially due to pain in deeper structures such as internal organs, joints, muscles or bones
3. Inability to participate in the study, in the opinion of the investigator, because of, for example, severe brain damage, language barrier, dementia, or other clinically significant or unstable conditions
4. Subjects using adjuvant chemotherapy or radiotherapy; adjuvant therapies must have been finished at least 4 weeks prior to the run-in period (Day -14)
5. Creatinine clearance <60 mL/min using the Cockcroft-Gault formula
6. White blood cell count <2500/mm³; neutrophil count <1500/mm³; platelet count <100 x 103/mm³
7. Heart rate <50 or >100 beats per minute; systolic blood pressure <100 or >140 mmHg; diastolic blood pressure <50 or >90 mmHg after 5 minutes rest in supine position
8. A history of multiple drug allergies
9. History or presence of alcohol or drug abuse
10. Subjects using strong opioids (e.g. a Morphine Equivalent Dose [MED] >80 mg/day)
11. Positive test for drugs of abuse at Day -7
12. Evidence of depression and/or a score of ≥11 on the HADS depression subscale
13. Any clinically relevant psychiatric disease in the past 5 years which is likely to interfere with the conduct of the study
14. History of any clinically relevant liver disease within the last 6 months, or episodic/chronic migraine, or kidney dysfunction or disease
15. Clinically significant gastrointestinal conditions, likely interfering with the study medication, study procedures or the outcome of the study
16. Positive test for human immunodeficiency virus (HIV)
17. Positive test for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C antibody and/or HIV1/HIV2 antibody at Screening
18. Participation of subject in an interventional clinical study within 1 month or, if applicable, 5 half-lives of the IMP, whatever is longer, before Screening or during participation in this study
19. Subjects who were previously enrolled in this clinical study and have taken study medication or terminated due to poor compliance
20. Known hypersensitivity to the active substance or any of the excipients of the IMP or the rescue medication
21. Subjects dependent (as an employee or relative) on the sponsor or investigator
22. Subjects committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
23. Legal incapacity or limited legal capacity

Randomization criteria

1. At least 5 daily pain assessments in the baseline week prior to randomization, with a mean score on the PI-NRS ≥4 and ≤9. Differences between the baseline daily pain scores on the PI-NRS must be ≤50%.
2. For female subjects of childbearing potential: negative pregnancy test in urine on Day 1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Day 10 in the 5-day average pain intensity score based on the Pain Intensity Numerical Rating Scale (PI-NRS; ranges from "no pain" = 0 to "the worst possible pain" = 10; the lower the score, the better the outcome) | Baseline to Day 10
  The 5-day average pain intensity score based on the Pain Intensity Numerical Rating Scale (PI-NRS) will be assessed to investigate the efficacy of repeat oral dosing of AP-325

SECONDARY OUTCOMES:
Longitudinal analysis of the 5-day average PI-NRS score (ranges from "no pain" = 0 to "the worst possible pain" = 10; the lower the score, the better the outcome) over time from Baseline until Day 35 | Baseline to Day 35
  The 5-day average PI-NRS score will be assessed to investigate the long-lasting efficacy of repeat oral dosing of AP-325 on neuropathic pain over the entire study duration
Changes from Baseline in the 5-day average PI-NRS score (change can be in the range of 0 to 10; the bigger the change towards lower PI-NRS scores, the better the outcome) (from Baseline to Day 5, 15, 20, 25, 30 and 35) | Baseline to Day 5, 15, 20, 25, 30 and 35
  The 5-day average PI-NRS score will be assessed
Responder rate: proportion of subjects who have a ≥30% reduction in the 5-day average PI-NRS score (in the range of 0 to 10; the bigger the change towards lower scores, the better the outcome) relative to Baseline (on Days 5, 10, 15, 25 and 35) | Baseline to Day 5, 10, 15, 25 and 35
  The responder rate will be compared between treatments on Day 5, 10, 15, 25 and 35
Responder rate: proportion of subjects who have a ≥50% reduction in the 5-day average PI-NRS score (in the range of 0 to 10; the bigger the change towards lower scores, the better the outcome) relative to Baseline (on Days 5, 10, 15, 25 and 35) | Baseline to Day 5, 10, 15, 25 and 35
  The responder rate will be compared between treatments on Day 5, 10, 15, 25 and 35
Proportion of subjects who "much improved" or "very much improved" relative to Baseline on the patient global impression of change (PGIC) on Days 3, 10, 15, and 36 | Days 3, 10, 15, and 36
  The PGIC will be dichotomized into treatment success (i.e. scoring 'much improved' or 'very much improved').
Changes from Baseline in the neuropathic pain evaluation using the neuropathic pain symptom inventory (NPSI; ranges from "no pain" = 0 to "the worst possible pain" = 120; the lower the score, the better) questionnaire on Days 3, 10, 15, and 36 | Baseline, Day 3, 10, 15 and 36
  Neuropathic pain symptom inventory (NPSI) questionnaire to assess the neuropathic pain of the patients
Changes from Baseline in the 5-day average daily sleep interference scale (DSIS; ranges from "pain does not interfere with sleep" = 0 to "pain completely interferes with sleep" = 10) score (from Baseline to Day 5, 10, 15, 25 and 35) | Baseline to Day 5, 10, 15, 25 and 35
  The 5-day average daily sleep interference scale (DSIS) score will be assessed
Changes from Baseline in the anxiety and depression assessment using the hospital anxiety and depression scale (HADS; subscales range from 0 to 21, with higher values indicating higher anxiety or depression; the lower the score) on Days 10 and 36 | Baseline, Day 10 and 36
  The hospital anxiety and depression scale (HADS) to assess the anxiety and depression of the patients
Time to first use of rescue medication after randomization | A priori specification not possible, between Day 1 until Day 36
  The time to first use of rescue medication after randomization will be analyzed
Total amount of rescue medication use (in mg per day) after randomization | A priori specification not possible, between Day 1 until Day 36
  The total amount of rescue medication (i.e. the total mg of rescue medication per day will be tabulated
Proportion of subjects classified as treatment failure | A priori specification not possible, between Day1 and Day 36
  Proportion of subjects classified as treatment failure at least once after randomization will be tabulated
Time to classification as treatment failure after randomization | A priori specification not possible, between Day1 and Day 36
  Time to first classification as treatment failure after randomization will be analyzed
Incidence, severity and seriousness of treatment-emergent adverse events (TEAEs) | A priori specification not possible, between Day1 and Day 36
  All TEAEs occurring during the clinical trial will be registered, documented and evaluated
Incidence of abnormal physical examinations | Baseline, Day 3, 10, 15 and 36
  Abnormal physical examination results will be evaluated and reported as AEs
Changes from Baseline in vital signs: Systolic and diastolic blood pressure | Baseline, Day 1, 3, 10, 15 and 36
  Systolic and diastolic blood pressure will be measured
Changes from Baseline in vital signs: Heart rate | Baseline, Day 1, 3, 10, 15 and 36
  Heart rate will be measured
Changes from Baseline in vital signs: Respiratory rate | Baseline, Day 1, 3, 10, 15 and 36
  Respiratory rate will be measured
Changes from Baseline in vital signs: Aural body temperature | Baseline, Day 1, 3, 10, 15 and 36
  Aural body temperature will be measured
Incidence of abnormal laboratory test results | Baseline, Day 3, 10, 15 and 36
  Abnormal laboratory test results will be evaluated
Incidence of abnormal ECG readings | Baseline, Day 3, 10 and 36
  Abnormal 12 lead ECG readings will be evaluated
Changes from Baseline in body weight | Baseline, Day 10 and 36
  Body weight will be evaluated
Plasma concentrations of AP-325 at 1 hour post-dose on Days 1 and 10; pre-dose on Days 3 and 10; and on Day 36 | Days 1, 3, 10 and 36
  Plasma concentrations of AP-325 will be evaluated
Accumulation of Ctrough from Day 3 to Day 10 | Day 3 and 10
  Plasma concentrations of AP-325 will be evaluated
Correlation between Ctrough-ss (Day 10) and the change from Baseline to Day 10 in the 5-day average pain intensity score based on the PI-NRS | Baseline to Day 10
  AP-325 concentration-effect relationships will be evaluated
Correlation between CYP2C9 genotype and the metabolism of AP-325 (optional) | Day 3
  The effect of CYP2C9 polymorphisms (determined by CYP2C9 genotyping) on the plasma concentration of AP-325 will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Heike Rittner, Prof. Dr., Principal Investigator — Universitätsklinikum Würzburg, Interdisziplinäre Schmerzmedizin, Germany
Locations (32):
- Belgium (6):
  - UZ Antwerp, Edegem
  - Ziekenhuis Oost Limburg - campus St. Jan, Genk
  - AZ Sint-Lucas, Pijnkliniek, Ghent
  - Jessa ZH Hospital, Hasselt
  - UZ Leuven, Campus Pellenberg, Pellenberg
  - AZ Delta, Pijncentrum, Roeselare
- Czechia (6):
  - Neurology and Physiotherapy Outpatient Clinic Skopalíkova, Brno
  - NEUROHK, s.r.o., Choceň
  - ALGOMED s.r.o. - Centrum léčby bolesti, České Budějovice
  - Neuros, s.r.o., Pilsen
  - Praglandia, s.r.o., Prague
  - MP-neuro s.r.o., Poliklinika Modrý pavilon, Slezská Ostrava
- France (6):
  - CHU Amiens-Picardie, Centre de Recherche Clinique, Amiens
  - Institut de Cancerologie de l'Ouest, Anesthésie/Douleur, Angers
  - Hopital Ambroise Paré, Centre d'évaluation et de traitement de la douleur, Boulogne
  - CHD Vendée, Département d'évaluation et du traitement de la douleur, La Roche-sur-Yon
  - Polyclinique de Limoges - Site Chenieux, Centre d'Evaluation et de traitement de la Douleur, Limoges
  - Hopîtal Cochin, Centre d'évaluation et du traitement de la douleur, Paris
- Germany (5):
  - emovis GmbH, Dedicated Study Site, Berlin
  - Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil gGmbH, (Ruhr-Universität Bochum) Neurologische Klinik und Poliklinik, Bochum
  - Kliniken der Stadt Köln gGmbH, Krankenhaus Köln-Merheim, Lungenklinik am Zentrum für Thoraxchirurgie, Pneumologie/ Onkologie, Schlaf- und Beatmungsmedizin, Klinikum der Universität Witten/Herdecke, Cologne
  - Florence-Nightingale-Krankenhaus der Kaiserswerther Diakonie, Klinik für Thoraxchirurgie, Düsseldorf
  - Universitätsklinikum Würzburg, Klinik und Poliklinik für Anästhesiologie, Zentrum für Interdisziplinäre Schmerzmedizin, Würzburg
- Spain (9):
  - HOSPITAL DEL MAR.#Cod. CNH: 080057#, Barcelona
  - HOSPITAL UNIVERSITARIO PUERTA DEL MAR#Cod. CNH: 110012#, Cadiz
  - HOSPITAL UNIVERSITARI DE BELLVITGE#Cod. CNH: 080752#, L'Hospitalet de Llobregat
  - HOSPITAL UNIVERSITARIO 12 DE OCTUBRE#Cod. CNH: 280035#, Madrid
  - HOSPITAL UNIVERSITARIO LA PAZ#Cod. CNH: 280014#, Madrid
  - HOSPITAL UNIVERSITARIO LA MORALEJA#Cod. CNH: 281179#, Madrid
  - CLINICA UNIVERSIDAD DE NAVARRA#Cod. CNH: 310060#, Pamplona
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID#Cod. CNH: 281203#, Pozuelo de Alarcón
  - HOSPITAL CLINICO UNIVERSITARIO DE VALENCIA#Cod. CNH: 460044#, Valencia

IPD SHARING:
Plan to Share IPD: No